CLINICAL TRIAL: NCT03196479
Title: Comparison Between Efficacy of Ketamine and Propofol Mixture With 1:6 Ratio and 1:4 Ratio for Endoscopic Retrograde Procedure Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Rudyanto Sedono, Anesthesiology Consultant, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes017
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Adult Patients Undergoing ERCP
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketamine:propofol ratio of 1:6 (Active Comparator): K16 group was received ketamine:propofol with ratio of 1:6, filled in 50 cc syringe, which consisted of 1 ml of ketamine (50 mg/ml), 30 ml of 1% propofol (10 mg/ml), and 19 ml of normal saline so that every ml of mixture consisted of 1 mg of ketamine and 6 mg of propofol
  Interventions: Drug: ketamine and propofol mixture with 1:6 ratio
- ketamine:propofol ratio of 1:4 (Active Comparator): K14 group was received ketamine:propofol with ratio of 1:4, filled in 50 cc syringe, which consisted of 1 ml of ketamine (50 mg/ml), 20 ml of 1% propofol (10 mg/ml), and 29 ml of normal saline so that every ml of mixture consisted of 1 mg of ketamine and 4 mg of propofol
  Interventions: Drug: ketamine and propofol mixture with 1:4 ratio

INTERVENTIONS:
Drug: ketamine and propofol mixture with 1:6 ratio — K16: K16 group was received ketamine:propofol with ratio of 1:6, filled in 50 cc syringe, which consisted of 1 ml of ketamine (50 mg/ml), 30 ml of 1% propofol (10 mg/ml), and 19 ml of normal saline so that every ml of mixture consisted of 1 mg of ketamine and 6 mg of propofol
  Arms: ketamine:propofol ratio of 1:6
Drug: ketamine and propofol mixture with 1:4 ratio — K14 group was received ketamine:propofol with ratio of 1:4, filled in 50 cc syringe, which consisted of 1 ml of ketamine (50 mg/ml), 20 ml of 1% propofol (10 mg/ml), and 29 ml of normal saline so that every ml of mixture consisted of 1 mg of ketamine and 4 mg of propofol
  Arms: ketamine:propofol ratio of 1:4

SUMMARY:
This study aimed to compare the efficacy of ketamine and propofol mixture with 1:6 ratio and 1:4 ratio for endoscopic retrograde procedure

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine Universitas Indonesia was acquired prior conducting the study. Subjects were given informed consent before enrolling the study. Intravenous (IV) cannula (20 G) , non-invasive blood pressure monitor, and pulse-oxymetry had been set on the subjects in endoscopic room. Vital signs were recorded. Subjects were then randomized into two groups (Ketamine:propofol ratio of 1:6 [K16] and ketamine:propofol ratio of 1:4 [K14]). K16 group's drug mixture was ketamine:propofol with ratio of 1:6, filled in 50 cc syringe, which consisted of 1 ml of ketamine (50 mg/ml), 30 ml of 1% propofol (10 mg/ml), and 19 ml of normal saline so that every ml of mixture consisted of 1 mg of ketamine and 6 mg of propofol. K14 group's drug mixture was ketamine:propofol with ratio of 1:4, filled in 50 cc syringe, which consisted of 1 ml of ketamine (50 mg/ml), 20 ml of 1% propofol (10 mg/ml), and 29 ml of normal saline so that every ml of mixture consisted of 1 mg of ketamine and 4 mg of propofol. Patient then was given initial bolus dose of 1 mg/kg body weight (BW) (based on propofol dose) and continued with maintenance dose of propofol (50 mcg/kg BW/minute, based on propofol dose). Maintenance dose could be increased by 10 mcg/kg BW/ minute if the subject still gave response to surgical stimulation or decreased by 10 mcg/kg BW/minute if hypotension occured. Onset of the drug, vital signs every 5 minutes, hypotension and desaturation events were recorded. If there were signs of pain such as tachycardia or hypertension, an additional dose of 25 mcg of fentanyl intravenous was given and recorded. After the endoscopic retrograde cholangiopancreatography (ERCP) finished, drugs were stopped and the total doses of propofol, drug administration speed, total dose of fentanyl used, and recovery time were recorded. Subjects were moved to the recovery room and observed for side effects event. Subjects were moved to the ward after aldrete score of 9-10.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were going to undergo ERCP unders sedation. Patient with American Society of Anesthesiologists (ASA) physical status of I-III, and body mass index of 18-30 kg/m2.

Exclusion Criteria:

* Subjects with history of allergy with drugs used in this trial, subjects with cardiovascular disease, hypertension, respiratory disorder, pregnancy, unstable hemodynamic, psychiatric drugs consumption, possibility of difficult airway, and kidney disorder

Drop out Criteria:

* drug allergy during procedure, hypotension (>20%) not resolved using ephedrine, desaturation (oxygen saturation <90%) not resolved using positive pressure ventilation, and endoscopic complication occur

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Recovery Time | Day 1
  Recovery time after procedure has ended
Propofol requirement | Day 1
  Total dose of propofol used during ERCP
Fentanyl requirement | Day 1
  Total dose of fentanyl used during ERCP

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Central Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ASGE Standards of Practice Committee; Early DS, Ben-Menachem T, Decker GA, Evans JA, Fanelli RD, Fisher DA, Fukami N, Hwang JH, Jain R, Jue TL, Khan KM, Malpas PM, Maple JT, Sharaf RS, Dominitz JA, Cash BD. Appropriate use of GI endoscopy. Gastrointest Endosc. 2012 Jun;75(6):1127-31. doi: 10.1016/j.gie.2012.01.011. No abstract available. PMID 22624807
- [Background] Triantafillidis JK, Merikas E, Nikolakis D, Papalois AE. Sedation in gastrointestinal endoscopy: current issues. World J Gastroenterol. 2013 Jan 28;19(4):463-81. doi: 10.3748/wjg.v19.i4.463. PMID 23382625
- [Background] Nwokediuko SC, Obienu O. Sedation practices for routine diagnostic upper gastrointestinal endoscopy in Nigeria. World J Gastrointest Endosc. 2012 Jun 16;4(6):260-5. doi: 10.4253/wjge.v4.i6.260. PMID 22720128
- [Background] Andolfatto G, Willman E. A prospective case series of pediatric procedural sedation and analgesia in the emergency department using single-syringe ketamine-propofol combination (ketofol). Acad Emerg Med. 2010 Feb;17(2):194-201. doi: 10.1111/j.1553-2712.2009.00646.x. PMID 20370749
- [Background] Goudra BG, Singh PM. Propofol alternatives in gastrointestinal endoscopy anesthesia. Saudi J Anaesth. 2014 Oct;8(4):540-5. doi: 10.4103/1658-354X.140893. PMID 25422614
- [Background] Sharieff GQ, Trocinski DR, Kanegaye JT, Fisher B, Harley JR. Ketamine-propofol combination sedation for fracture reduction in the pediatric emergency department. Pediatr Emerg Care. 2007 Dec;23(12):881-4. doi: 10.1097/pec.0b013e31815c9df6. PMID 18091596
- [Background] Kogan A, Efrat R, Katz J, Vidne BA. Propofol-ketamine mixture for anesthesia in pediatric patients undergoing cardiac catheterization. J Cardiothorac Vasc Anesth. 2003 Dec;17(6):691-3. doi: 10.1053/j.jvca.2003.09.008. PMID 14689406
- [Background] Botero CA, Smith CE, Holbrook C, Chavez AM, Snow NJ, Hagen JF, Pinchak AC. Total intravenous anesthesia with a propofol-ketamine combination during coronary artery surgery. J Cardiothorac Vasc Anesth. 2000 Aug;14(4):409-15. doi: 10.1053/jcan.2000.7933. PMID 10972606
- [Background] Coulter FL, Hannam JA, Anderson BJ. Ketofol simulations for dosing in pediatric anesthesia. Paediatr Anaesth. 2014 Aug;24(8):806-12. doi: 10.1111/pan.12386. Epub 2014 Mar 26. PMID 24666723
- See also: Glomsaker TB. Endoscopic Retrograde Cholangiopancreatography (ERCP) in Norway. University of Bergen, 2013. — http://bora.uib.no/handle/1956/7581
- See also: Donnelly RF, Willman E, Andolfatto G. Stability of Ketamine - Propofol Mixtures for Procedural Sedation and Analgesia in the Emergency Department. Can J Hosp Pharm 2008; 61: 426-430. — http://www.cjhp-online.ca/index.php/cjhp/article/view/99
- See also: Wang Y. A randomized double-blind controlled study of the efficacy of ketofol with propofol-fentanyl and propofol alone in termination of pregnancy. African J Pharm Pharmacol 2012; 6: 2510-2514. — http://www.academicjournals.org/journal/AJPP/article-abstract/CCEDA2F29373